CLINICAL TRIAL: NCT01122979
Title: National (Brazil), Phase IV, Multicentric, Open Label, Parallel, Comparative Study of the Use of Insulin Glargine + Glulisine or Insulin Regular + NPH Insulin (Isophane Insulin) in Type 2 Diabetes Mellitus Patients With Moderate Renal Failure.
Brief Title: Evaluation of the Safety and Efficacy of Insulin Glargine + Glulisine or Insulin Regular + NPH Insulin (Isophane Insulin) Use in Type 2 Diabetes Mellitus Patients With Moderate Renal Failure.
Acronym: DINAMO
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Sanofi (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: LANTU_L_04737
Record Dates: First submitted 2010-05-11; First posted 2010-05-13 (Estimated); Last update posted 2013-11-08 (Estimated); Status verified 2013-11

CONDITIONS: Diabetes Mellitus, Type 2
MeSH Terms: conditions — Diabetes Mellitus, Type 2 | interventions — Insulin Glargine; Insulin, Isophane; insulin glulisine; Insulin

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- group 1: insulin glargine + insulin glulisine (Experimental): insulin glargine once daily + glulisine at meal times
  Interventions: Drug: INSULIN GLARGINE; Drug: INSULIN GLULISINE
- group 2 NPH insulin + regular insulin (Active Comparator): NPH insulin (isophane insulin) (2 or more divided doses) + regular insulin at meal times
  Interventions: Drug: NPH insulin (insulin isophane); Drug: Regular insulin

INTERVENTIONS:
Drug: INSULIN GLARGINE — Pharmaceutical form: 100 Units/mL solution for injection in a pre-filled SoloStar pen (3 mL) Route of administration: subcutaneous Dose regimen: dose adjusted to the patient's glycemia
  Arms: group 1: insulin glargine + insulin glulisine
Drug: NPH insulin (insulin isophane) — Pharmaceutical form: solution for injection Route of administration: subcutaneous Dose regimen: dose adjusted to the patient's glycemia
  Arms: group 2 NPH insulin + regular insulin
Drug: INSULIN GLULISINE — Pharmaceutical form: 100 Units/mL solution for injection in a pre-filled SoloStar pen (3 mL) Route of administration: subcutaneous Dose regimen: dose adjusted to the patient's glycemia
  Arms: group 1: insulin glargine + insulin glulisine
Drug: Regular insulin — Pharmaceutical form: solution for injection Route of administration: subcutaneous Dose regimen: dose adjusted to the patient's glycemia
  Arms: group 2 NPH insulin + regular insulin

SUMMARY:
Primary Objective:

>To obtain an estimation for both treatment groups of the proportion of patients that reach the target of HbA1c <= 7% without confirmed nocturnal hypoglycaemia in each treatment group.

Secondary Objectives:

* Glycemic control, measured by HbA1c and FPG (fasting plasma glucose) at baseline and after each period of treatment.
* Incidence of confirmed symptomatic and nocturnal hypoglycemia.
* Incidence of confirmed severe hypoglycemia (< 36mg/dL or need of help to recover). >Weight variation for each period of treatment.
* Creatinine clearance at baseline and after each period of treatment.
* Overall safety: Incidence of adverse events.

ELIGIBILITY:
Inclusion criteria:

* Type 2 diabetes and renal failure in use of NPH regular insulin or fast-acting analog and HbA1c >= 8%.
* Albuminuria or microalbuminuria diabetic retinopathy.
* Creatinine clearance < 60 mL/min/1,73 m2 and >30 mL/min/1,73 m2

Exclusion criteria:

* Hypersensibility to insulin glargine or any other component of the insulin formulation.
* Use of investigational medications during the last 12 months or use of any investigational insulin preparation during the last 4 months.
* History of diabetic ketoacidosis or positive GAD antibodies.
* Advanced retinopathy needing laser therapy.
* Diagnosed advanced neuropathy
* Severe hepatic disease or active hepatitis.
* Cardiac failure class III or IV (NYHA).
* Patients on hemodialysis.
* Diagnosed cancer.
* Active infection.
* Current therapy with steroids.
* Patients with recognized or suspected endocrine disorders associated with increased insulin resistance, acromegaly, or hyperthyroidism.

The above information is not intended to contain all considerations relevant to a patient's potential participation in a clinical trial.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 72 (Actual)
Dates: Start 2010-07; Primary Completion 2013-10 (Actual); Study Completion 2013-10 (Actual)

PRIMARY OUTCOMES:
Proportion of patients that reach the target of HbA1c ≤7% without confirmed nocturnal hypoglycaemia in each treatment group and the respective CI 90%. | From visit 1 (Day 1) to visit 13 (Day 169)

SECONDARY OUTCOMES:
Proportion of patients that reach the target of HbA1c ≤7% and proportion of patients reaching the target of Fasting Plasma Glucose (FPG ≤100mg/dL). | From baseline and Visit 13 (Day 169)
Incidence of confirmed symptomatic and nocturnal hypoglycemias: plasma glucose measurement <= 70mg/dL. | From baseline and Visit 13 (Day 169)
Incidence of confirmed severe hypoglycemia: plasma glucose level < 36 mg/dL (2 mmol/L) or with prompt recovery after oral carbohydrate, intravenous glucose, or glucagon administration | From baseline and Visit 13 (Day 169)
Weight variation | From baseline to the end of treatment at visit 13 (day 169)
Creatinine clearance variation | From baseline to the end of treatment at visit 13 (day 169)

CONTACTS AND LOCATIONS:
Overall Officials: Clinical Sciences & Operations, Study Director — Sanofi
Locations (10):
- Brazil (10):
  - Investigational Site Number 076-007, Curitiba
  - Investigational Site Number 076-010, Fortaleza
  - Investigational Site Number 076-001, Fortaleza
  - Investigational Site Number 076-003, Porto Alegre
  - Investigational Site Number 076-005, São Paulo
  - Investigational Site Number 076-013, São Paulo
  - Investigational Site Number 076-004, São Paulo
  - Investigational Site Number 076-002, São Paulo
  - Investigational Site Number 076-009, São Paulo
  - Investigational Site Number 076-006, Taguatinga